CLINICAL TRIAL: NCT07258472
Title: Multidimensional Assessment of Preoperative Anxiety and Quality of Life on Postoperative Patient-Reported Outcomes Following Free Gingival Graft Surgery
Brief Title: Impact of Preoperative Anxiety on Postoperative Quality of Life After Free Gingival Graft Surgery
Acronym: FGG-QoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Collaborators: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Serap Karakış Akcan, Assistant professor doctor, DDS, PhD, Istanbul Gelisim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: B.30.2.AYD.0.00.00-480.2/130
Record Dates: First submitted 2025-09-04; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Gingival Recession; Dental Anxiety; Quality of Life
Keywords: free gingival graft; Oral Health-Related Quality of Life (OHRQoL); State-Trait Anxiety Inventory (STAI); Patient-Reported Outcomes
MeSH Terms: conditions — Gingival Recession | interventions — fibrinopeptides gamma; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Single-arm interventional study in which all participants undergo free gingival graft surgery and are evaluated for preoperative anxiety, postoperative pain, and quality of life outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Free Gingival Graft (FGG) Surgery (Experimental): All participants underwent free gingival graft (FGG) surgery using a standardized protocol performed by the same surgical team. Local anesthesia was administered, a half-thickness flap was prepared, and grafts harvested from the palatal donor site were secured with sutures. Postoperative care included analgesics and chlorhexidine mouth rinse. Sutures and periodontal dressing were removed at day 14.
  Interventions: Procedure: Free Gingival Graft (FGG) Surgery

INTERVENTIONS:
Procedure: Free Gingival Graft (FGG) Surgery

SUMMARY:
This study investigates the effect of free gingival graft (FGG) surgery on patients' oral health-related quality of life (QoL) during the first postoperative month and evaluates the role of preoperative anxiety on postoperative QoL outcomes. Thirty-six participants indicated for FGG surgery due to insufficient keratinized gingiva were included. The Oral Health Impact Profile-14 (OHIP-14) was administered preoperatively, daily during the first postoperative week, and at one month. Preoperative anxiety levels were assessed using the State-Trait Anxiety Inventory (STAI-S and STAI-T). Postoperative pain was evaluated with the Visual Analog Scale (VAS) for seven days. Demographic and lifestyle variables, including age, gender, educational status, marital status, and smoking status, were recorded. Clinical parameters such as plaque and gingival indices and keratinized tissue width were measured preoperatively and one month postoperatively. Intraoperative surgical data, including graft vertical height, horizontal width, thickness, and recipient site dimensions, were documented. Statistical analysis will determine the relationship between preoperative anxiety and postoperative QoL, as well as the influence of surgical and demographic factors on patient-reported outcomes.

DETAILED DESCRIPTION:
Free gingival graft (FGG) procedures are widely used to increase keratinized gingiva and manage mucogingival problems. Despite predictable clinical outcomes, these surgeries are associated with postoperative discomfort, donor site morbidity, and aesthetic limitations that may negatively affect patient quality of life (QoL). Preoperative anxiety is also considered an important factor influencing postoperative pain perception and recovery.

This prospective clinical study was conducted between August 2016 and May 2017 to evaluate the effect of FGG surgery on oral health-related quality of life (OHQoL) and to investigate the relationship between preoperative anxiety and postoperative outcomes. Thirty-six participants who met the eligibility criteria underwent FGG surgery following phase I periodontal therapy.

Preoperative assessments included demographic data, plaque index, gingival index, keratinized tissue width, and anxiety levels measured using the State-Trait Anxiety Inventory (STAI-S and STAI-T). The OHIP-14 questionnaire was completed one week before surgery, on the day of surgery, daily for the first seven postoperative days, and at one month.

Intraoperative variables recorded included graft vertical height, horizontal width, thickness, and recipient site dimensions. Postoperative assessments included OHIP-14 scores, Visual Analog Scale (VAS) scores for pain collected daily for seven days, the number of analgesics used, and clinical measurements of gingival indices and keratinized tissue width at one month.

The primary outcome is the change in OHIP-14 scores over time and their association with preoperative anxiety. Secondary outcomes include postoperative pain, analgesic consumption, and the influence of surgical and demographic parameters on QoL.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years

Systemically healthy

Non-smokers or smoking fewer than 10 cigarettes per day

Healthy periodontal and peri-implant tissues

Presence of ≤2 teeth or implants in the recipient area with keratinized tissue width (KTW) < 1 mm

Not pregnant or lactating

No bleeding disorders

Not taking medications that could interfere with wound healing

Provided complete responses to all follow-up questionnaires

* Exclusion Criteria:

Previous history of periodontal surgical treatment

Difficulty reading or understanding the questionnaires

Failure to follow the study timeline (e.g., missed or late responses)

Presence of active periapical or peri-implant infection at the surgical site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change in Oral Health Impact Profile-14 (OHIP-14) Total Score | Baseline, Day 1-7, and 1 month after surgery
  Oral health-related quality of life will be evaluated using the Oral Health Impact Profile-14 (OHIP-14), as derived and validated by Slade (1997, Community Dent Oral Epidemiol, 25: 284-90). Each of the 14 items is scored on a 0-5 scale (0 = never, 5 = very often), producing a total score ranging from 0 to 70. Higher scores indicate poorer oral health-related quality of life. Changes in total OHIP-14 scores will be recorded from baseline to postoperative Day 1-7 and 1 month.
  Unit of Measure:
  Score (0-70)
Correlation Between Preoperative Anxiety Levels (STAI-S and STAI-T) and Postoperative OHIP-14 Score Changes | Baseline and 1 month after surgery
  Correlation between changes in Oral Health Impact Profile-14 (OHIP-14) scores and preoperative anxiety levels will be evaluated using the State-Trait Anxiety Inventory (STAI-S for state anxiety and STAI-T for trait anxiety). Each STAI subscale ranges from 20 to 80, with higher scores indicating greater anxiety. Correlation analysis (Pearson's r or Spearman's ρ) will be performed to determine whether baseline anxiety levels are associated with postoperative changes in OHIP-14 total scores.
  Unit of Measure:
  Correlation coefficient (r)

SECONDARY OUTCOMES:
Correlation Between OHIP-14 Scores and Demographic and Surgical Factors | Baseline, Day 1-7, and 1 month after surgery
  Correlation analyses will be performed to evaluate the relationship between postoperative OHIP-14 total scores and demographic (age, gender, education, marital status, smoking status) and surgical factors (graft dimensions, recipient site dimensions, operation duration).
  Unit of Measure:
  Correlation coefficient (r)
Postoperative Pain Intensity (VAS) | Day 1-7 after surgery
  Postoperative pain intensity will be assessed daily during the first postoperative week using a 100-mm Visual Analog Scale (VAS), where 0 represents no pain and 100 represents the worst imaginable pain. Higher scores indicate greater pain intensity.
  Unit of Measure:
  Score (0-100 mm)
Analgesic Consumption During the First Postoperative Week | Day 1-7 after surgery
  Participants recorded the number of analgesic tablets taken each day during the first postoperative week. Total analgesic consumption will be calculated as the sum of doses taken over 7 days.
  Unit of Measure:
  Number of tablets per week
Plaque Index Score (Silness-Löe) | Baseline and 1 month postoperatively
  Plaque Index (Silness-Löe) scores will be recorded at baseline and 1 month after surgery to evaluate plaque accumulation around the treated sites. Each surface is scored from 0 to 3, where 0 indicates no plaque and 3 indicates abundant soft deposits. Higher scores indicate greater plaque accumulation.
  Unit of Measure:
  Score (0-3)
Gingival Index Score (Löe-Silness) | Baseline and 1 month postoperatively
  Gingival Index (Löe-Silness) scores will be recorded at baseline and 1 month after surgery to evaluate gingival inflammation around the treated sites. Each surface is scored from 0 to 3, where 0 indicates normal gingiva and 3 indicates severe inflammation with ulceration or spontaneous bleeding. Higher scores indicate more severe gingival inflammation.
  Unit of Measure:
  Score (0-3)
Keratinized Tissue Width (mm) | Baseline and 1 month postoperatively.
  Description:
  The width of keratinized tissue will be measured in millimeters using a periodontal probe from the gingival margin to the mucogingival junction at baseline and 1 month after free gingival graft surgery.
  Unit of Measure:
  Millimeters (mm)

OTHER OUTCOMES:
Graft Dimensions (Vertical Height and Horizontal Width) | At surgery (baseline)
  The vertical height (GVH) and horizontal width (GHW) of the free gingival graft will be measured in millimeters during surgery using a manual caliper. The graft vertical height will be recorded as the apico-coronal dimension, and the horizontal width as the mesio-distal dimension of the harvested graft.
  Unit of Measure:
  Millimeters (mm)
Graft Thickness (GT) | At surgery (baseline)
  Description:
  The graft thickness will be measured in millimeters using a manual caliper at the mid-point of the harvested graft during surgery.
  Unit of Measure:
  Millimeters (mm)
Recipient Site Dimensions (Horizontal Width and Vertical Depth) | At surgery (baseline)
  The recipient site horizontal width (RHW) will be measured as the widest mesio-distal distance, and the recipient site vertical depth (RVD) as the deepest apico-coronal distance, using a manual caliper during surgery.
  Unit of Measure:
  Millimeters (mm)
Surgery Duration | At surgery
  The duration of surgery will be recorded in minutes, measured from the first incision until placement of the final suture using a stopwatch.
  Unit of Measure:
  Minutes (min)

CONTACTS AND LOCATIONS:
Overall Officials: serap karakış akcan, DDS,PhD, Principal Investigator — stanbul Gelişim University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Istanbul Gelisim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Zucchelli G, Tavelli L, McGuire MK, Rasperini G, Feinberg SE, Wang HL, Giannobile WV. Autogenous soft tissue grafting for periodontal and peri-implant plastic surgical reconstruction. J Periodontol. 2020 Jan;91(1):9-16. doi: 10.1002/JPER.19-0350. Epub 2019 Oct 6. PMID 31461778
- [Result] Bitencourt FV, Cardoso De David S, Schutz JDS, Otto Kirst Neto A, Visioli F, Fiorini T. Minimizing patient morbidity after free gingival graft harvesting:A triple-blind randomized-controlled clinical trial. Clin Oral Implants Res. 2022 Jun;33(6):622-633. doi: 10.1111/clr.13923. Epub 2022 Apr 6. PMID 35305280
- [Result] Mounssif I, Bentivogli V, Rendon A, Gissi DB, Maiani F, Mazzotti C, Mele M, Sangiorgi M, Zucchelli G, Stefanini M. Patient-reported outcome measures after periodontal surgery. Clin Oral Investig. 2023 Dec;27(12):7715-7724. doi: 10.1007/s00784-023-05362-y. Epub 2023 Nov 9. PMID 37940683
- [Result] Zucchelli G, Mounssif I, Mazzotti C, Montebugnoli L, Sangiorgi M, Mele M, Stefanini M. Does the dimension of the graft influence patient morbidity and root coverage outcomes? A randomized controlled clinical trial. J Clin Periodontol. 2014 Jul;41(7):708-16. doi: 10.1111/jcpe.12256. Epub 2014 May 8. PMID 24708394
- [Result] Ozcelik O, Haytac MC, Seydaoglu G. Immediate post-operative effects of different periodontal treatment modalities on oral health-related quality of life: a randomized clinical trial. J Clin Periodontol. 2007 Sep;34(9):788-96. doi: 10.1111/j.1600-051X.2007.01120.x. PMID 17716314
- [Result] Fardal O, McCulloch CA. Impact of anxiety on pain perception associated with periodontal and implant surgery in a private practice. J Periodontol. 2012 Sep;83(9):1079-85. doi: 10.1902/jop.2011.110562. Epub 2011 Dec 19. PMID 22181682
- [Result] Croog SH, Baume RM, Nalbandian J. Pre-surgery psychological characteristics, pain response, and activities impairment in female patients with repeated periodontal surgery. J Psychosom Res. 1995 Jan;39(1):39-51. doi: 10.1016/0022-3999(94)00089-n. PMID 7760302
- [Result] McGrath C, Bedi R. The association between dental anxiety and oral health-related quality of life in Britain. Community Dent Oral Epidemiol. 2004 Feb;32(1):67-72. doi: 10.1111/j.1600-0528.2004.00119.x. PMID 14961842
- [Result] Sen DO, Sengul BI, Yarkac FU, Oncu E. Impact of platelet-rich fibrin derivatives on patient morbidity and quality of life in palatal donor sites following free gingival graft surgery: a randomized clinical trial. Clin Oral Investig. 2024 Nov 7;28(12):631. doi: 10.1007/s00784-024-06023-4. PMID 39505777